CLINICAL TRIAL: NCT06863922
Title: A Pilot Study of Berberine (Soloways ™) in Patients with Type 2 Diabetes Mellitus Carrying TCF7L2 Polymorphisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW020
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; type 2 diabetes; supplements; genetics; berberine; HbA1c
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCF7L2 Homozygous Variant Cohort (Experimental)
  Interventions: Dietary Supplement: Berberine
- Non-Variant (Control) Cohort (Active Comparator)
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Dietary Supplement: Berberine — Berberine 500-1000 mg, administered 2-3 times per day for 12 weeks, in addition to standard of care
  Arms: Non-Variant (Control) Cohort
Dietary Supplement: Berberine — Berberine 500-1000 mg, administered 2-3 times per day for 12 weeks, in addition to standard of care
  Arms: TCF7L2 Homozygous Variant Cohort

SUMMARY:
This pilot, genotype-stratified clinical trial aims to investigate the safety and preliminary efficacy of berberine supplementation in adult patients with type 2 diabetes mellitus (T2DM) who carry a specific high-risk TCF7L2 polymorphism (e.g., rs7903146) in the homozygous state. The study will compare improvements in glycemic control and metabolic markers between two groups: (1) homozygous carriers of the TCF7L2 "unfavorable" variant and (2) non-carriers (wild-type). It is hypothesized that berberine will yield greater reductions in HbA1c and fasting plasma glucose among homozygous carriers, potentially due to their distinct TCF7L2-mediated insulin secretion and sensitivity pathways.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is driven by a combination of insulin resistance and impaired insulin secretion. Genetic polymorphisms in the transcription factor 7-like 2 (TCF7L2) gene have been strongly associated with an increased risk of T2DM, potentially through altered beta-cell function and incretin signaling. Berberine, a natural alkaloid derived from plants such as Coptis chinensis, has demonstrated hypoglycemic effects by modulating pathways like AMPK, thereby improving insulin sensitivity and glucose metabolism. This pilot trial aims to clarify whether berberine offers a more pronounced metabolic benefit to individuals homozygous for a "high-risk" TCF7L2 polymorphism by targeting their unique pathophysiological mechanisms. Results will inform future larger-scale, genotype-focused interventional trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 30-70 years) with a confirmed diagnosis of type 2 diabetes mellitus.
* On stable doses of metformin or other standard oral antihyperglycemic agents for at least 4 weeks prior to enrollment.
* Willingness to undergo genetic testing for TCF7L2 polymorphisms. For the Homozygous Variant Cohort: confirmed homozygous high-risk TCF7L2 polymorphism (e.g., rs7903146) prior to enrollment.
* For the Non-Variant Cohort: confirmed wild-type TCF7L2 genotype.

Exclusion Criteria:

* Current use of insulin therapy or recent (within 4 weeks) change in diabetic medications.

Known hypersensitivity or intolerance to berberine or related compounds.

* Significant renal or hepatic impairment.
* Pregnancy or breastfeeding.
* Any other acute or chronic condition that, in the investigator's judgment, could compromise the patient's safety or the study's integrity.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) | 12 weeks
Change in Fasting Plasma Glucose (FPG) | 12 weeks

SECONDARY OUTCOMES:
Change in HOMA-IR (Insulin Resistance Index) | 12 weeks
Number of Adverse Events | 12 weeks
Change in Lipid Profile Triglyceride | 12 weeks
Change in Lipid Profile LDL-C | 12 weeks
Change in Lipid Profile HDL-C | 12 weeks
Change in Body Weight or Body Mass Index (BMI) | 12 weeks
Change in Patient-Reported Quality of Life as Measured by the World Health Organization | 12 weeks
  Patient-reported quality of life will be assessed using the World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF). This validated questionnaire provides scores ranging from 0 to 100 for each domain (physical health, psychological health, social relationships, and environment), where higher scores indicate a better quality of life. The outcome will be reported as the mean change in the relevant domain scores from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No